CLINICAL TRIAL: NCT03646565
Title: A Longitudinal Study and Follow-up of the Psychosocial Development and Investigation of the Wellbeing of Children Undergoing Open Cardiac Surgery in Their Early Ages.
Brief Title: Psychosocial Development of Children Undergoing Open Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Semmelweis University Heart and Vascular Center (Other)
Responsible Party: Sponsor
Other Study IDs: ChildrenHeart
Record Dates: First submitted 2018-08-23; First posted 2018-08-24 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Cardiac Surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In recent years, improvement of medical treatments leads to the effect, that 90% of children originally born with congenital heart disease (CHD) are reaching adulthood. Mortality rates have significantly decreased in the last decades. However several studies have shown that with multiple consequences have to face the survivors. Eg. neuronal and psychological injuries during the perioperative period. After all, the surgical interventions that save their lives might result in psychological and behavioral deviations and increased morbidity, which is strongly worsening the quality of life, learning abilities and behavioral development of these patients. Not yet available any clinical guidelines for managing or screening these patients for designing intervention, taking corrective actions.

The investigators wish to identify those perioperative factors that might affect the well-being, coping, the behavior alteration and psychosocial status of children, who underwent open chest cardiac interventions in early ages. The investigators also wish to understand the long-term changes of the illness-representation of this population and to see its effect for the wellbeing and coping.

DETAILED DESCRIPTION:
The study population will include school-aged children treated and followed in the Gottsegen György Hungarian Institute of Cardiology in Budapest. The participants will be selected from patients who underwent open-chest cardiac surgery, under the age of four, between 2003- 2007 and once followed up in 2013-2014.

Psychosocial measures will be as follows: Beck Depression Inventory (BDI), Spielberger State-Trait Anxiety Inventory (STAI-S/T), KidScreen questionnaire, PRISM-D and person/organ test.

A range of perioperative and psychosocial factors will be assessed as potential determinants of outcome. The data will be fully retrieved from the registries of our hospital center. Characteristics registered included pre-, intra- and postoperative variables such as age, gender, comorbidities (renal, hepatic, infectious, neurological, metabolic, hormonal or genetic disorders), type of surgery, laboratory parameters, operation time, cardiopulmonary bypass (CPB) time, aortic cross-clamp time, Risk Assessment for Congenital Heart Surgery (RACHS) points, length of mechanical ventilation, blood loss, transfusions, fluid balance, need for inotropic support or pulmonary vasodilatation, medications, anaesthetic and analgesic agents.

By comparing the above mentioned perioperative data with the result of the psychological measures we expect to answer our hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent open-chest heart surgery between 2003-2007
* Operated patients (surgery made between 2003-2007) who had been followed up by the institution between 2013-14. and filled in the psychological questionnaires

Exclusion Criteria:

- Patients who had not been followed up by the institution between 2013-14 and thus had not filled the psychological questionnaires

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population included school-aged children treated and followed in the Gottsegen György Hungarian Institute of Cardiology in Budapest. The operated subgroup enrolled patients who underwent open chest cardiac surgery, under the age of four, between 2003-2007
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Well-being measured with the KidScreen52 questionnaire | 11-15 years after the intervention
  Items scored on a 5-point scale ranging from never / not at all to always. 10 dimensions (no. of items)
  * Physical- (5) Max. score (MS) = higher physically fit, active, healthy.
  * Psychological Well-being (6). MS = more happy, views life positively, satisfied.
  * Moods and Emotions (7). MS: more good feelings, good mood.
  * Self-Perception (5). MS: higher level of self-confident, positive body image.
  * Autonomy (5). MS: is feels free to decide, independent, autonomous.
  * Parent Relations and Home Life (6). MS: feels secure, supported and loved.
  * Social Support and Peers (6). MS: feels accepted, supported and included in peer group.
  * School Environment (6). MS: feels happy at school and doing well.
  * Social Acceptance (Bullying) (3). MS: not feeling bullied, feeling respected and accepted by peers.
  * Financial Resources (3). MS: higher security in terms of financial resources.
Illness representation measured with PRISM-D and person/organ test | 11-15 years after the intervention
  PRISM-D; person/organ test: both used for illness representation. Patients is given to a landscape oriented a4 white paper with a yellow circle on the left down corner. The Investigator ask the patient to imagine that the white paper his/her life and the yellow circle is him/herself. Than patient instructed to first draw another circle with red that represent him/her illness. Than the investigator asks him/her to draw all the people and things important to him/her at this very moment in his life by using different colors. Scored based on the distance, size, etc.
  According to the person/organ test' instruction the patient first have to draw him/herself, than his/her heart. Based on the location of the organ, and it's distance from the body scoring is made.

CONTACTS AND LOCATIONS:
Locations (1):
- Semmelweis University, Budapest, Hungary